CLINICAL TRIAL: NCT00340366
Title: Investigation Into the Influence of Genetic Variation on Folate, Cobalamin and Related Metabolites
Brief Title: Influence of Genetics on Vitamin Metabolism in Pregnant Women
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904068; 04-HG-N068
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-10

CONDITIONS: Pregnancy; Birth Defects
Keywords: Homocysteine; Vitamin B12; Birth Defects; Pregnancy; Folate; Irish Individuals
MeSH Terms: conditions — Congenital Abnormalities

SUMMARY:
This study will examine how the body metabolizes micronutrients, such vitamins, during pregnancy and how genetic make-up influences their metabolism. Vitamin B12 and folate levels in pregnancy have been linked to birth defects, such as neural tube defects, orofacial clefts, and congenital heart disease. Other micronutrient levels may be related to other birth defects or pregnancy complications. This study will characterize the patterns of micronutrient status during pregnancy and compare it with genetic variants and biochemical parameters. Information about the relationship between genes and vitamin metabolism may help doctors advise women about their nutritional requirements during pregnancy to protect their health and the health of their babies.

This study is a collaboration between NIH and Trinity College in Dublin, Ireland. Women of Irish origin 18 years of age or older who are receiving prenatal care at the Coombe Women's Hospital in Dublin may be enrolled. Fathers also may participate.

Upon entering the study, female participants complete a questionnaire relating to their food and vitamin intake, alcohol consumption, smoking behavior, and use of medications, and provide a blood sample. Additional blood samples are collected during routine clinic visits at about 24 and 34 weeks of pregnancy, and again at delivery and from 6 weeks to 2 months after the baby's birth. Permission will be requested to obtain a blood sample from the umbilical cord at birth after it has been removed from the baby.

Fathers of the babies are also asked to answer a short questionnaire and to provide a DNA sample for genetic studies. To collect the DNA, sterile cotton swabs are rubbed around the inside of the mouth to obtain cheek cells from which the DNA is extracted.

DETAILED DESCRIPTION:
A number of genetic polymorphisms influence human folate, vitamin B12 and related micronutrient levels. Vitamin B12 and folate levels in pregnancy have been linked to birth defects including neural tube defects, orofacial clefts, and congenital heart disease. Additionally, related analytes, such as homocysteine, may be related to birth defects and pregnancy complications. The behavior of maternal serum micronutrients and related analytes throughout human pregnancy is not well described. In this study, we aim to characterize the patterns of micronutrient status during pregnancy. We plan to perform biochemical analyses on serial blood samples collected from 500 pregnant women at five intervals spanning early pregnancy and the post partum period. We will also characterize neonatal micronutrient status using a specimen of umbilical cord blood. These blood specimens, as well as buccal swab specimens collected from the fathers, will also be evaluated to measure the influence of genetic variants on metabolite levels. The major outcomes measured will be longitudinal maternal micronutrient levels and aggregate alleel frequencies among family triads. Comparisons will be made between the presence of genetic variants, biochemical parameters, and clinical phenotype. At a later date we also plan to study the same metabolic and genetic parameters in a large cohort of healthy individuals. Characterizing these biochemical and genetic variants should provide insight into the metabolic processes of normal and complicated pregnancies.

ELIGIBILITY:
* Eligible participants will be women of Irish origin (older than 18) presenting for prenatal care to the Coombe Women's Hospital, Dublin, Republic of Ireland. Non-Irish women (a small proportion of the population) will be excluded because the prevalence of genetic polymorphisms can vary greatly among different populations; we already have an estimate of the distribution of this genotype in the Irish women. Members of the only minority group native to Ireland, the Travelers, will not be excluded. While culturally distinct, the Travelers are genetically similar to the majority population. Women with multiple pregnancy (more than one fetus) and users of IV drugs will be excluded. Women will be asked for permission to obtain a cord blood sample from the infant at delivery. Women will be asked to assist with recruitment of their partners (father of the fetus), who will be included if they consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2003-12-16; Study Completion 2007-12-10

CONTACTS AND LOCATIONS:
Locations (1):
- The Coombe Maternity Hospital, Dublin, Ireland

REFERENCES:
- [Background] Kirke PN, Molloy AM, Daly LE, Burke H, Weir DG, Scott JM. Maternal plasma folate and vitamin B12 are independent risk factors for neural tube defects. Q J Med. 1993 Nov;86(11):703-8. PMID 8265769